CLINICAL TRIAL: NCT03692416
Title: The Effect of Some Drugs Used in Treatment of Vasculitis on the Complement System in Children Attending Assiut University Hospital.
Brief Title: The Effect of Some Drugs Used in Treatment of Vasculitis on the Complement System in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RIHassan, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANCA
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Vasculitis
Keywords: C3,C4, C5a & ANCA
MeSH Terms: conditions — Vasculitis | interventions — Ibuprofen; Prednisone; Methotrexate

STUDY DESIGN:
Intervention Model Description: The aim of this work is to assess the effect of various forms of treatment of vasculitis on C3, C4, C5a & ANCA levels in blood, in infants & children.
Masking Description: No other parties are masked in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen (Active Comparator): Patients in this group will receive:
  Ibuprofen
  * Oral
  * At a dosage of 30 to 40 mg/kg/day, divided into 3 or 4 doses/day, max 2400 mg/day, given with food, in the form of suspension or tablets.
  * Duration of therapy: 4 - 6 weeks.
  Interventions: Drug: Ibuprofen
- Prednisone Oral or Methylprednisolone IV (Active Comparator): Steroids:
  1. Pednisone (for mild/moderate cases):
     * Oral
     * Single daily morning dosage of 0.05-2.0 mg/kg/day, or in 2 - 4 divided doses, max 80 mg/d.
     * Duration: 4 - 6 weeks, with gradual tapering to the lowest effective dose.
  2. Methylprednisolone (for severe/acute cases):
     * IV
     * 10-30 mg/kg/dose (max 1 g), over 1 hr daily for 1-5 days, followed by oral prednisone, with gradual tapering to the lowest effective dose.
     * The duration is variable according to the condition of the patient.
  Interventions: Drug: Prednisone
- Methotrexate (Active Comparator): Patients in this group will receive:
  Methotrexate
  * Oral
  * At a dosage of 10 to 20 mg/m2/wk (0.35 to 0.65 mg/kg/wk), max dose 25 mg/wk.
  * Duration of therapy: 6 - 12 weeks.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Ibuprofen — Infants and children with vasculitis attending AssiutU, aged > 1 mo. - 17 yr. of both genders will be included during 2 years of study.
  Besides full clinical history and thorough examination, all cases will have: CBC, CRP, ESR, Renal function tests & Albumin / creatinine ratio.
  All cases will have an initial estimation as well as follow up estimation after treatment by Ibuprofen for ANCA, C3, C4 &C5a levels done, measured By ELISA technique.
  Other Names: Advil
  Arms: Ibuprofen
Drug: Prednisone — Infants and children with vasculitis attending AssiutU, aged > 1 mo. - 17 yr. of both genders will be included during 2 years of study.
  Besides full clinical history and thorough examination, all cases will have: CBC, CRP, ESR, Renal function tests & Albumin / creatinine ratio.
  All cases will have an initial estimation as well as follow up estimation after treatment by Steroids for ANCA, C3, C4 &C5a levels done, measured By ELISA technique.
  Other Names: Deltasone Oral or Solu-Medrol IV
  Arms: Prednisone Oral or Methylprednisolone IV
Drug: Methotrexate — Infants and children with vasculitis attending AssiutU, aged > 1 mo. - 17 yr. of both genders will be included during 2 years of study.
  Besides full clinical history and thorough examination, all cases will have: CBC, CRP, ESR, Renal function tests & Albumin / creatinine ratio.
  All cases will have an initial estimation as well as follow up estimation after treatment by Methotrexate for ANCA, C3, C4 &C5a levels done, measured By ELISA technique.
  Other Names: Rheumatrex
  Arms: Methotrexate

SUMMARY:
Vasculitis denotes affection of small to medium sized vessels by polyangitis. Antineutrophil cytoplasmic antibodies (ANCA) are immunoglobulin G (IgG) autoantibodies directed against constituents of neutrophil granules leading to neutrophil degeneration which results in cell apoptosis known as "Natoptosis" (NaTosis) of the cells. These lead to vessel endothelial cell damage. So that, ANCA formation seems to be the basic reaction in vasculitis.

Complement activation at C3 and C4 was thought to be involved in renal damage ANCA associated vasculitis (AAV).

DETAILED DESCRIPTION:
Vasculitis syndromes include: Henoch-Schonlein Purpura (HSP), connective tissue disorders e.g. Systemic Lupus Erythematosus (SLE), Rheumatoid arthritis...etc; where small vessels are mainly involved in the process of vasculitis. Vasculitis syndromes also include Kawasaki disease where also medium sized vessels are also included. Other vasculitis syndromes are also reported.

ANCA associated vasculitis may be due complex interplay of genetic risks, environmental or infection trigger or adaptive immunity leading to insufficient regulation of B cells with pathogenic ANCA generation and neutrophil activation (AAV).

Complement activation at C3 and C4 was involved in organ damage, especially renal, in AAV at the alternative complement pathway, factor B and properdin component colocalized with C3 complement in the endothelium of the blood vessels.

Furthermore, the common complement pathway was activated as reflected by increased C5a levels. This suggests that both the alternative and common complement pathways are involved in some cases of vasculitis. Furthermore a decrease in these activation factors was observed during remission of vasculitis. This may denote clearance of the degradation of cell component that were blocking inactive vasculitis. In addition, many studies noticed strong increased plasma levels of the anaphlatoxin C5a that has a strong proinflammatory activity on the endothelium of vessels that may be related to disease severity. So much so, that inhibition of C5a levels by immunologic inhibitors may have a therapeutic role in some forms of ANCA positive vasculitis.

Various treatment forms have been used for vasculitis syndromes.

* Drugs used in treatment of Juvenile Idiopathic Arthritis (JIA) are:

  1. Non-steroidal Anti-inflammatory Drugs (NSAIDs) such as Salicylates e.g. Aspirin, Selective COX-2 inhibitors e.g. Celecoxib & Non-Selective COX-2 inhibitors e.g. Naproxen.
  2. Non-biologic Disease-Modifying Anti-rheumatic drugs such as Methotrexate.
  3. Biologic Disease-Modifying Anti-rheumatic Drugs such as Infliximab.
  4. Oral or parenteral Glucocorticoids such as Methylprednisolone (According to American College of Rheumatology).
* In cases of SLE, the American College of Rheumatology (ACR) recommended corticosteroids in the 1st place and change to or add Biologic Disease-Modifying Anti-rheumatic Drugs Agents such as Rituximab.
* Regarding Henoch-Schonlein Purpura vasculitis, 70% of cases are self-limited. only cases with suspected renal involvement e.g. hematuria, hypertension, headache or proteinuria are to be treated with sreroids.

ELIGIBILITY:
Inclusion Criteria:

* Infants & children with vasculitis attending Assiut University Child Hospital (AUCH), aged > 1 mo. - 17yr. of both genders will be included during 2 years of study.

Exclusion Criteria:

* Those cases aged less than one month will be excluded from the study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2021-11-11 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
The serum levels of C3, C4 & C5a as an indicator of its therapeutic effect. | 2 years
  An initial estimation as well as follow up estimation after treatment for ANCA, C3, C4 &C5a levels done, measured By ELISA technique.

CONTACTS AND LOCATIONS:
Overall Officials: Safiea AF El-Deeb, PROF, Study Director — Assiut University Child Hospital
Locations (1):
- Assiut University Pediatric Hospital, Asyut, Upper Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting in January 2021
Access Criteria: through finding the research in the site of ClinicalTrials.gov
URL: http://rehabibrahem@gmail.com

REFERENCES:
- [Background] Chen SF, Wang FM, Li ZY, Yu F, Chen M, Zhao MH. The functional activities of complement factor H are impaired in patients with ANCA-positive vasculitis. Clin Immunol. 2017 Feb;175:41-50. doi: 10.1016/j.clim.2016.11.013. Epub 2016 Dec 6. PMID 27939215
- [Background] Gou SJ, Yuan J, Chen M, Yu F, Zhao MH. Circulating complement activation in patients with anti-neutrophil cytoplasmic antibody-associated vasculitis. Kidney Int. 2013 Jan;83(1):129-37. doi: 10.1038/ki.2012.313. Epub 2012 Aug 22. PMID 22913983
- [Background] Heineke MH, Ballering AV, Jamin A, Ben Mkaddem S, Monteiro RC, Van Egmond M. New insights in the pathogenesis of immunoglobulin A vasculitis (Henoch-Schonlein purpura). Autoimmun Rev. 2017 Dec;16(12):1246-1253. doi: 10.1016/j.autrev.2017.10.009. Epub 2017 Oct 14. PMID 29037908
- [Background] Jarrot PA, Kaplanski G. Pathogenesis of ANCA-associated vasculitis: An update. Autoimmun Rev. 2016 Jul;15(7):704-13. doi: 10.1016/j.autrev.2016.03.007. Epub 2016 Mar 9. PMID 26970490
- [Background] Kallenberg CG, Heeringa P. Complement is crucial in the pathogenesis of ANCA-associated vasculitis. Kidney Int. 2013 Jan;83(1):16-8. doi: 10.1038/ki.2012.371. PMID 23271485
- [Background] Noone D, Hebert D, Licht C. Pathogenesis and treatment of ANCA-associated vasculitis-a role for complement. Pediatr Nephrol. 2018 Jan;33(1):1-11. doi: 10.1007/s00467-016-3475-5. Epub 2016 Sep 5. PMID 27596099
- [Background] Pipitone N, Salvarani C. The role of infectious agents in the pathogenesis of vasculitis. Best Pract Res Clin Rheumatol. 2008 Oct;22(5):897-911. doi: 10.1016/j.berh.2008.09.009. PMID 19028370
- [Background] von Borstel A, Sanders JS, Rutgers A, Stegeman CA, Heeringa P, Abdulahad WH. Cellular immune regulation in the pathogenesis of ANCA-associated vasculitides. Autoimmun Rev. 2018 Apr;17(4):413-421. doi: 10.1016/j.autrev.2017.12.002. Epub 2018 Feb 9. PMID 29428808
- See also: Nelson Textbook of Pediatrics Expert Consult, Chapter 161, 1-8. — https://www.ClinicalGate.com/vasculitis-syndromes-2
- See also: American College of Rheumatology (ACR) Juvenile Idiopathic Arthritis Guideline Project Plan - June 2017 — https://www.rheumatology.org/Practice-Quality/Clinical-Support/Clinical-Practice-Guidelines/Rheumatoid-Arthritis